CLINICAL TRIAL: NCT04239976
Title: Effect of Scramble Therapy on Chemotherapy Induced Peripheral Neuropathic Pain: A Prospective, Pilot Study
Brief Title: Scrambler Therapy for the Reduction of Chemotherapy-Induced Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0651; NCI-2019-08323 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0651 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (scrambler therapy, sensory test, gait test) (Experimental): Patients undergo scrambler therapy over 30-45 minutes QD Monday-Friday for 2 weeks. Patients also undergo a quantitative sensory test and a gait assessment test using a FitBit before receiving scrambler therapy, at the end of the first and second weeks of scrambler therapy, and 1 month after the last day of scrambler therapy.
  Interventions: Device: FitBit; Other: Gait Assessment Test; Other: MC5-A Scrambler Therapy; Other: Quality-of-Life Assessment; Procedure: Quantitative Sensory Testing; Other: Questionnaire Administration

INTERVENTIONS:
Device: FitBit — Wear FitBit for gait assessment test
Other: Gait Assessment Test — Undergo gait assessment test
Other: MC5-A Scrambler Therapy — Undergo scrambler therapy
  Other Names: Scrambler Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Quantitative Sensory Testing — Undergo quantitative sensory test
  Other Names: QST
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well scrambler therapy works in reducing chemotherapy-induced neuropathic pain in patients with cancer. Scrambler therapy is a type of treatment that uses electrodes placed on the skin. Electricity is carried from the electrodes through the skin and blocks the pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of MC5-A scrambler therapy (scrambler therapy [ST]) in reducing chemotherapy-induced painful peripheral neuropathy (CIPPN).

II. Evaluate the change in pain score before and after 2 weeks (Monday-Friday) of the final ST treatment.

III. Assess for changes in other symptom burden (i.e insomnia, feeling of well-being, depression and anxiety) after 2 weeks (Monday-Friday) ST treatment.

SECONDARY OBJECTIVES:

I. To evaluate the following with the treatment of ST:

Ia. Assess for changes in therapy induced neuropathy assessment scale (TNAS). Ib. Assess for changes in using pain medications. Ic. Assess for changes in daily physical activities/functional status. Id. Assess for changes in quality of life using European Organization of Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) (chemotherapy induced peripheral neuropathy) chemotherapy-induced neuropathic pain (CIPN) 20 questionnaire.

Ie. Assess overall satisfaction with the ST treatment using Global Impression of Change questionnaire.

TERTIARY (EXPLORATORY) OBJECTIVE:

I. Determine the change in sensation after 2 weeks (Monday-Friday) of the final ST treatment.

OUTLINE:

Patients undergo scrambler therapy over 30-45 minutes once daily (QD) Monday-Friday for 2 weeks. Patients also undergo a quantitative sensory test and a gait assessment test using a FitBit before receiving scrambler therapy, at the end of the first and second weeks of scrambler therapy, and 1 month after the last day of scrambler therapy.

After completion of study, patients are followed up weekly for 3 weeks and at 4 weeks after the last day of scrambler therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cancer and suffer from CIPN for at least 3 months after the end of their last cancer chemotherapy
* Have average pain intensity of at least 4/10
* Be in stable clinical situation (no surgery, radiotherapy, hormone therapy, chemotherapy or other treatment scheduled) in the month following the enrollment)
* Can give a written informed consent

Exclusion Criteria:

* Pre-existence or history of seizure
* Pre-existence or history of peripheral neuropathy due to a cause different from neurotoxic chemotherapy (i.e. idiopathic peripheral neuropathy, diabetic neuropathy
* Pregnancy
* Present with pacemaker or implantable defibrillators
* Present or past psychotropic substances and alcohol dependence
* Inability to understand patients' information and informed consent
* Skin lesion at the electrode placement site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Chemotherapy induced peripheral neuropathic pain (CIPN) score difference | Baseline to the last day of 2-week treatment
  Will be assessed using descriptive statistics such as mean, standard deviation, median, range and confidence intervals. The t-test or Wilcoxon rank sum test and Fisher's exact test may be used to compare variables between patient groups. Correlation between two continuous measures may be assessed using Pearson or Spearman correlation. Other statistical methods may be utilized when appropriate. The Pain inventory is an assessment of pain level on a 11-point numeric rating scales (0=none to 10=worst).

SECONDARY OUTCOMES:
Change in therapy-induced neuropathy | Baseline to the last day of 2-week treatment
  Will be assessed using therapy induced neuropathy assessment scale. Will be assessed using descriptive statistics such as mean, standard deviation, median, range and confidence intervals. The t-test or Wilcoxon rank sum test and Fisher's exact test may be used to compare variables between patient groups. Correlation between two continuous measures may be assessed using Pearson or Spearman correlation. Other statistical methods may be utilized when appropriate.
Change in cancer-related symptoms | Baseline to the last day of 2-week treatment
  Will be assessed using therapy induced neuropathy assessment scale. Will be assessed using descriptive statistics such as mean, standard deviation, median, range and confidence intervals. The t-test or Wilcoxon rank sum test and Fisher's exact test may be used to compare variables between patient groups. Correlation between two continuous measures may be assessed using Pearson or Spearman correlation. Other statistical methods may be utilized when appropriate.
Change in physical function and quality of life | Baseline to the last day of 2-week treatment
  Will be assessed using the European Organization of Research and Treatment of Cancer Quality of Life Questionnaire CIPN20 questionnaire. Will be assessed using descriptive statistics such as mean, standard deviation, median, range and confidence intervals. The t-test or Wilcoxon rank sum test and Fisher's exact test may be used to compare variables between patient groups. Correlation between two continuous measures may be assessed using Pearson or Spearman correlation. Other statistical methods may be utilized when appropriate. The Pain inventory is an assessment of pain level on a 11-point numeric rating scales (0=none to 10=worst).

CONTACTS AND LOCATIONS:
Overall Officials: Salahadin Abdi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org